CLINICAL TRIAL: NCT01457209
Title: Effect of Acupuncture on Insulin Sensitivity in Women With and Without Polycystic Ovary Syndrome
Brief Title: Acupuncture to Treat Insulin Resistance in Women With and Without Polycystic Ovary Syndrome
Acronym: PCOS-AcupIR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCOS-AcupIR
Record Dates: First submitted 2011-10-06; First posted 2011-10-21 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Polycystic Ovary Syndrome; Insulin Resistance
Keywords: PCOS; Insulin resistance; Acupuncture
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Acupuncture — Needle placement in abdominal muscles, in m. vastus lateralis, lower leg and hands.
  Stimulation: Manual rotation of the needles and electrical stimulation of the needles in the abdominal muscles and m. vastus lateralis will be stimulated electrically with low burst frequency Duration: 30 min Treatment: 3 times/wk during 5 weeks.

SUMMARY:
The central hypothesis is that acupuncture break the vicious circle of androgen excess and reverse insulin resistance and improve health related quality of life and affective symptoms in overweight and obese women with and without Polycystic Ovary Syndrome.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is the most common endocrine and metabolic disorder in women. The main metabolic phenotype is hyperinsulinemia and insulin resistance, which are independent of body weight and worsen hyperandrogenism and ovulatory dysfunction. Pharmacological treatments are symptom oriented and usually effective but have metabolic and gastrointestinal side effects. Therefore, it is important to evaluate new nonpharmacological treatment strategies, as most women with PCOS require long-term treatment.

Hypothesis and Aims Our central hypothesis is that acupuncture break the vicious circle of androgen excess and reverse insulin resistance and improve health related quality of life and affective symptoms in overweight and obese women with and without PCOS.

The specific aim are designed to test the hypotheses that

1. Acupuncture (acute and chronic i.e. 5 weeks treatment, 3 times per week) improves insulin sensitivity in overweight and obese women with and without PCOS
2. Acupuncture (acute and chronic i.e. 5 weeks treatment, 3 times per week) regulate key signaling molecules and mitochondrial oxidation/biogenesis in skeletal muscle and adipose tissue in overweight and obese women with and without PCOS
3. Acupuncture (chronic i.e. 5 weeks treatment, 3 times per week) improve health related quality of life and symptoms of anxiety and depression in overweight and obese women with and without PCOS

Time frame of the study is 5-6 weeks. No long term follow up.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 25 to < 35 and
* Clinical signs of hyperandrogenism (hirsutism or acne) and
* At least one of the following two signs; oligo/amenorrhea and/or ultrasound-verified polycystic ovaries

Controls should have BMI > 25 to < 35, regular cycles with 28 days ± 2 days, no signs of hyperandrogenism.

Exclusion Criteria:

Exclusion criteria for all women

1. Age > 38 years
2. Exclusion of other endocrine disorders such as hyperprolactinemia (s-prolactin < 27µg/L), nonclassic congenital adrenal hyperplasia (17-hydroxyprogesterone < 3nmol/L), and androgen secreting tumors.
3. Autoimmune disorders, cancer, Type I diabetes and Type 2 diabetes.
4. Pharmacological treatment (cortisone, antidepressant, antidiabetic, hormonal contraceptives, hormonal ovulation induction or other drugs judged by discretion of investigator) within 12 wks accounts for all participants.
5. Blood pressure >160 / 100 mmHg
6. Pregnancy or breastfeeding the last 6 months
7. Acupuncture last 2 months
8. Language barrier or disabled person with reduced ability to understand information.

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2011-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in insulin sensitivity | Day 1 and Week 5
  glucose disposal rate measured by euglycemic hyperinsulinemic clamp.

SECONDARY OUTCOMES:
Change in insulin signaling (muscle and adipose tissue) | Day 1 and Week 5
  Western blot, RT-PCR
Change in health related quality of life | Day 1 and Week 5
  PCOSQ, SF36
Change in symptoms of anxiety and depression | Day 1 and Week 5
  CPRS-SA
Change in circulating sex steroids, adipokines, lipids and inflammatory markers | Day 1 and Week 5
  Mass spectrometry, ELISA

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Neuroscienncec and Physiology, Gothenburg, Sweden

REFERENCES:
- [Derived] Benrick A, Pillon NJ, Nilsson E, Lindgren E, Krook A, Ling C, Stener-Victorin E. Electroacupuncture Mimics Exercise-Induced Changes in Skeletal Muscle Gene Expression in Women With Polycystic Ovary Syndrome. J Clin Endocrinol Metab. 2020 Jun 1;105(6):2027-41. doi: 10.1210/clinem/dgaa165. PMID 32232327
- [Derived] Nilsson E, Benrick A, Kokosar M, Krook A, Lindgren E, Kallman T, Martis MM, Hojlund K, Ling C, Stener-Victorin E. Transcriptional and Epigenetic Changes Influencing Skeletal Muscle Metabolism in Women With Polycystic Ovary Syndrome. J Clin Endocrinol Metab. 2018 Dec 1;103(12):4465-4477. doi: 10.1210/jc.2018-00935. PMID 30113663
- [Derived] Zheng Y, Stener-Victorin E, Ng EH, Li J, Wu X, Ma H. How does acupuncture affect insulin sensitivity in women with polycystic ovary syndrome and insulin resistance? Study protocol of a prospective pilot study. BMJ Open. 2015 May 3;5(4):e007757. doi: 10.1136/bmjopen-2015-007757. PMID 25941189